CLINICAL TRIAL: NCT00312689
Title: Microbiological Examination of Children Operated for Congenital Lacrimal Stenosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Muenster (Other)
Other Study IDs: Record 1
Record Dates: First submitted 2006-04-07; First posted 2006-04-10 (Estimated); Last update posted 2007-04-12 (Estimated); Status verified 2007-04

CONDITIONS: Congenital Lacrimal Stenosis
Keywords: congenital; lacrimal; stenosis; bacteria; microbiological
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Children with congenital lacrimal stenosis are treated by probing and intubation of the lacrimal drainage system.

Hypothesis: Microbiological findings at the time of insertion and removal of the silicon intubation have an influence on the clinical outcome and success rate of the surgical treatment. Microbiological specimens are taken from conjunctiva and nasal mucosa during the two procedures under general anaesthesia and from the silicon tube after removal and examined for bacterial contamination.

DETAILED DESCRIPTION:
Children (age 0-14 years) with congenital lacrimal stenosis in whom probing and intubation of the lacrimal drainage system is indicated are included the study after informed written consent by their parents. Microbiological specimens are taken bilaterally from conjunctiva and nasal mucosa during the two procedures under general anaesthesia (insertion and removal of the silicon intubation) and from the silicon tube after removal. Specimens are examined for bacterial contamination. Microbiological findings are correlated with clinical data about the further clinical course and especially the success of the surgical treatment.

ELIGIBILITY:
Inclusion Criteria: age 0-14 years, congenital lacrimal stenosis, informed consent by the parents -

Exclusion Criteria: none

-

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120
Dates: Start 2006-03; Study Completion 2007-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Annette Kolck, MD, Principal Investigator — University Hospital Muenster
Locations (1):
- Augenklinik, Münster, Germany